CLINICAL TRIAL: NCT01936376
Title: A Prospective Observational Study to Evaluate Acute Kidney Injury Biomarkers In Patients Receiving First Cycle of Cisplatin Chemotherapy for Head and Neck Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Foundation for the National Institutes of Health (Other)
Collaborators: University of Southern California (Other); University of Minnesota (Other); M.D. Anderson Cancer Center (Other); Brigham and Women's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Amgen (Industry); AstraZeneca (Industry); Eli Lilly and Company (Industry); Johnson & Johnson (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Critical Path Institute - Predictive Safety Testing Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: Kidney Safety - Cisplatin
Record Dates: First submitted 2013-08-29; First posted 2013-09-06 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Cancer
Keywords: kidney safety; biomarkers; serum creatinine; BUN; cystic fibrosis; head and neck cancer; renal injury; drug induced acute kidney injury; aminoglycoside; cisplatin; nephrotoxicity; biomarker qualification
MeSH Terms: conditions — Head and Neck Neoplasms; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- head & neck cancer patients, cisplatin treatment
- cancer patients, no cisplatin, no nephrotoxic agent

SUMMARY:
The project is designed to test new biomarkers that are more sensitive than the current standard in detecting injury to the proximal kidney tubule and will establish better criteria for when kidney safety concerns may halt further testing of a drug in humans.

DETAILED DESCRIPTION:
The study will be conducted at four major medical centers, including the University of Southern California, the University of Minnesota, the Dana Farber Cancer Institute, and the MD Anderson Cancer Center. Blood and urine samples will be collected from patients undergoing treatment with either cisplatin or aminoglycosides, which are two different drugs known to cause injuries to the proximal tubule of the kidney. Cisplatin is a common chemotherapy drug taken by patients with head and neck cancer. Aminoglycosides are a common antibiotic drug taken by patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria (Cisplatin Treatment Group):

1. Males and females ≥ 18 years of age
2. Diagnosis of head & neck cancer and confirmation that patient is due to receive a 1st cycle of cisplatin (75-100 mg/m2/cycle) chemotherapy either:

   * as single agent chemotherapy in conjunction with local radiotherapy course, or
   * as part of the TPF combination (docetaxel, cisplatin, and fluorouracil)
3. Willingness and ability to comply with study procedures and study restrictions
4. Ability to provide written informed consent

Inclusion Criteria (Control Group):

1. Males and females ≥ 18 years of age
2. Diagnosis of head & neck cancer or similar condition such as an upper body, localised malignancy. These control patients will be scheduled to receive a non-nephrotoxic treatment modality (e.g. local radiotherapy alone)
3. Willingness and ability to comply with study procedures and study restrictions
4. Ability to provide written informed consent

Exclusion Criteria (All Subjects):

1. Chronic kidney disease defined by eGFR <60 mL/min/1.73m2. Patients with normal eGFR but persistent dipstick proteinuria require urinary albumin measurement: those with microalbuminuria (>30 mcg/mg creatinine) will be excluded
2. Patients currently receiving other potentially nephrotoxic agents (i.e. chronic use of high dose NSAIDs, intravenous aminoglycosides, intravenous colistin, intravenous vancomycin, or ACEi)
3. Any major surgery (i.e. high risk of acute kidney injury) in the previous month
4. Patients currently receiving trimethoprim or cimetidine or other medications known to alter the tubular secretion of creatinine
5. Use of creatine supplements within 7 days prior to hospitalization
6. Solid organ transplant recipients
7. Abnormal liver function (serum ALT, AST or total bilirubin >2xULN)
8. Significant anemia (Hemoglobin < 10 g/dL)
9. Pregnancy
10. Institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
biomarker change from baseline | up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abdulla Salahudeen, MD, Principal Investigator — M.D. Anderson Cancer Center; Sushrut Waikar, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Harvard Medical School - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Texas MD Anderson, Houston, Texas